CLINICAL TRIAL: NCT02159859
Title: Pharmacokinetics and Investigation of Optimal Dose of Invanz (Ertapenem) in Hemodialysis Patients
Brief Title: Pharmacokinetics and Optimal Dose of Ertapenem in Hemodialysis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Corewell Health East (Other)
Collaborators: Wayne State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OH-D-Ertapenem-HD
Record Dates: First submitted 2014-06-03; First posted 2014-06-10 (Estimated); Results first posted 2017-06-15 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-09

CONDITIONS: End Stage Renal Disease
Keywords: ertapenem; pharmacokinetic; pharmacodynamics; hemodialysis; requires hemodialysis three times a week
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Ertapenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ertapenem (Experimental): Subjects with end stage renal disease (ESRD) who undergo hemodialysis three times a week and without infection will be administered one gram of ertapenem once over five minutes through infusion access after a hemodialysis session, and will have blood drawn at time 0, 0.5, 1, 2, 6, and 12 hours after the ertapenem administration and once prior to the next hemodialysis session
  Interventions: Drug: Ertapenem

INTERVENTIONS:
Drug: Ertapenem — Subjects are hemodialysis patients who are admitted to Oakwood Hospital - Dearborn
  Other Names: Invanz

SUMMARY:
The purpose of this study is to determine the amount of ertapenem in the blood over time between hemodialysis session.

DETAILED DESCRIPTION:
After a hemodialysis session, subject will be administered ertapenem and the amount of ertapenem in the blood will be measured at seven time periods before the initiation of the next hemodialysis session.

ELIGIBILITY:
Inclusion Criteria:

* Men or women age between 18 and 88 at the time of admission to Oakwood Hospital and Medical Center during January 1, 2014 or date of Institutional Review Board (IRB) approval to December 1, 2015
* Diagnosed with end stage renal disease and requires hemodialysis three times a week
* No allergy to β lactam medications
* Existing IV access for parenteral ertapenem infusion
* Willing for blood draws, at predose, 0.5, 1, 2, 6, 12 hours post-hemodialysis and pre-hemodialysis for the following hemodialysis and immediately post hemodialysis session and 1 hour post.
* No evidence of hepatic disease
* No history of alcoholism or drug abuse within pervious 2 years
* Not pregnant

Exclusion Criteria:

* History of any form of epilepsy, seizure or convulsion
* Currently taking any forms of valproic acid or divalproex sodium for treatment of any disease states
* Currently taking probenecid
* Current Clostridium difficile (C. diff.) infection, defined as 30 days prior to day-1 of receiving ertapenem for this study
* Currently receiving any antimicrobial agents for prophylaxis or treatment

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-12; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lama Hsaiky, Pharm.D., Principal Investigator — Oakwood Hospital - Dearborn; Lama Hsaiky, Pharm.D., Study Chair — Oakwood Hospital - Dearborn
Locations (1):
- Oakwood Hospital - Dearborn, Dearborn, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hsaiky LM, Salinitri FD, Wong J, Jennings ST, Desai NH, Lobkovich AM, Cha R. Pharmacokinetics and investigation of optimal dose ertapenem in intermittent hemodialysis patients. Nephrol Dial Transplant. 2019 Oct 1;34(10):1766-1772. doi: 10.1093/ndt/gfy166. PMID 29992286

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ertapenem
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Ertapenem: Pharmacokinetics and Optimal Dose of Ertapenem in Hemodialysis Patients
Arm/Group | Ertapenem
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7
weight [Mean (Standard Deviation); unit: kilograms] | 77.7 (18.3)

OUTCOME MEASURES:

1. Primary Outcome: Mean Maximum Concentration (Cmax) of Ertapenem in Hemodialysis Patients
Description: Mean Cmax will be calculated from a series of ertapenem concentration from the blood samples, i.e.once after hemodialysis session prior to ertapenem administration, and at 0.5, 1, 2, 6, 12 hours after the administration of one gram ertapenem over five minutes, and once before the next hemodialysis session
Time Frame: once after hemodialysis session prior to ertapenem administration and at 0.5, 1, 2, 6, 12 hours after the administration of one gram ertapenem over five minutes, and once before the next hemodialysis session
Measure: Mean (Standard Deviation); unit: mcg/ml
Arm/Group | Ertapenem
Number analyzed (Participants) | 7
mcg/ml | 663.1 (904.9)

2. Primary Outcome: Mean Minimum Concentration (Cmin) of Ertapenem in Hemodialysis Patients
Description: Mean Cmin will be calculated from a series of ertapenem concentration from the blood samples, i.e.once after hemodialysis session prior to ertapenem administration, and at 0.5, 1, 2, 6, 12 hours after the administration of one gram ertapenem over five minutes, and once before the next hemodialysis session
Time Frame: once after hemodialysis session prior to ertapenem administration, and at 0.5, 1, 2, 6, 12 hours after the administration of one gram ertapenem over five minutes, and once before the next hemodialysis session
Measure: Mean (Standard Deviation); unit: mcg/ml
Arm/Group | Ertapenem
Number analyzed (Participants) | 7
mcg/ml | 44.3 (14.5)

3. Primary Outcome: Mean Area Under the Curve (AUC) of Ertapenem in Hemodialysis Patients
Description: Mean AUC will be calculated from a series of ertapenem concentration from the blood samples, i.e.once after hemodialysis session prior to ertapenem administration, and at 0.5, 1, 2, 6, 12 hours after the administration of one gram ertapenem over five minutes, and once before the next hemodialysis session
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*ug/mL
Arm/Group | Ertapenem
Number analyzed (Participants) | 7
h*ug/mL | 6225 (1259)

4. Primary Outcome: Mean Terminal Half Life (t1/2) of Ertpenem in Hemodialysis Patients
Description: Mean t1/2 will be calculated from a series of ertapenem concentration from the blood samples, i.e.once after hemodialysis session prior to ertapenem administration, and at 0.5, 1, 2, 6, 12 hours after the administration of one gram ertapenem over five minutes, and once before the next hemodialysis session
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ertapenem
Number analyzed (Participants) | 7
hours | 19.3 (6.6)

5. Primary Outcome: Mean Time to Cmax of Ertapenem in Hemodialysis Patients
Description: Mean time to Cmax will be calculated from a series of ertapenem concentration from the blood samples, i.e.once after hemodialysis session prior to ertapenem administration, and at 0.5, 1, 2, 6, 12 hours after the administration of one gram ertapenem over five minutes, and once before the next hemodialysis session
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ertapenem
Number analyzed (Participants) | 7
hours | 0.5 (0)

6. Secondary Outcome: Number of Participants With Diarrhea
Description: Evaluation of diarrhea will be performed by the study physician at screening, predose, 24 hours, and 5 to 7 days after the ertapenem dose or the last day of patient's stay in the hospital
Time Frame: Up to seven days after the administration of ertapenem
Measure: Count of Participants; unit: Participants
Arm/Group | Ertapenem
Number analyzed (Participants) | 7
Participants | 1

7. Secondary Outcome: Number of Participants With Nausea and Vomiting
Description: Evaluation of nausea and vomiting will be performed by the study physician at screening, predose, 24 hours, and 5 to 7 days after the ertapenem dose or the last day of patient's stay in the hospital
Time Frame: Up to seven days after the administration of ertapenem
Measure: Count of Participants; unit: Participants
Arm/Group | Ertapenem
Number analyzed (Participants) | 7
Participants | 1

8. Secondary Outcome: Number of Participants With Headache
Description: Evaluation of headache will be performed by the study physician at screening, predose, 24 hours, and 5 to 7 days after the ertapenem dose or the last day of patient's stay in the hospital
Time Frame: Up to seven days after the administration of ertapenem
Measure: Count of Participants; unit: Participants
Arm/Group | Ertapenem
Number analyzed (Participants) | 7
Participants | 0

9. Secondary Outcome: Number of Participants With Injection Site Reaction
Description: Evaluation of injection site reaction will be performed by the study physician at screening, predose, 24 hours, and 5 to 7 days after the ertapenem dose or the last day of patient's stay in the hospital
Time Frame: Up to seven days after the administration of ertapenem
Measure: Count of Participants; unit: Participants
Arm/Group | Ertapenem
Number analyzed (Participants) | 7
Participants | 0

10. Other Pre Specified Outcome: Number of Participants With Any Adverse Events
Description: Evaluation of any adverse events will be performed by the study physician at screening, predose, 24 hours, and 5 to 7 days after the ertapenem dose or the last day of patient's stay in the hospital
Time Frame: Up to seven days after the administration of ertapenem
Measure: Count of Participants; unit: Participants
Arm/Group | Ertapenem
Number analyzed (Participants) | 7
Participants | 6

ADVERSE EVENTS:
Time Frame: within 7days post enrollment
Arm/Group | Ertapenem
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 6/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ertapenem (N=7)
hypoglycemia (Endocrine disorders) | 3 (3)
hypertension (Vascular disorders) | 2 (2)
nausea (Gastrointestinal disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Muscle jerking (Musculoskeletal and connective tissue disorders) | 1 (1)
Rusty urine (Renal and urinary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
some participants had missing lab values at the pre-determined times

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes